CLINICAL TRIAL: NCT03554031
Title: A Single Arm, Multicenter Phase III Clinical Trial to Evaluate the Efficacy and Safety of Recombinant Human Growth Hormone Injection in Patients With Prader-Willi Syndrome
Brief Title: A Study to Evaluate the Efficacy and Safety of Recombinant Human Growth Hormone Injection in Patients With Prader-Willi Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Children's Hospital of Fudan University (Other); Tongji medical college huazhong university of science & technology (Unknown); Beijing Children's Hospital (Other); Peking University First Hospital (Other); Peking Union Medical College Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci PWS CT
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rhGH injection/Jintropin AQ (Experimental): Drug: Recombinant Human Growth Hormone Injection /Jintropin AQ, 30IU/10 mg/3ml/kit, 0.5 mg/m2/d for the first 4 weeks, then 1.0 mg/m2/d for subsequent 48 weeks; by subcutaneous injection, once per day for total 52 weeks.No control.
  Interventions: Drug: Recombinant Human Growth Hormone (rhGH) Injection

INTERVENTIONS:
Drug: Recombinant Human Growth Hormone (rhGH) Injection — Drug: Recombinant Human Growth Hormone Injection /Jintropin AQ, 30IU/10 mg/3ml/kit, 0.5 mg/m2/d for the first 4 weeks, then 1.0 mg/m2/d for subsequent 48 weeks; by subcutaneous injection, once per day for total 52 weeks.

SUMMARY:
To evaluate the effectiveness of rhGH (Recombinant human growth hormone) injection for improving motor development in patients with PWS.

ELIGIBILITY:
Inclusion Criteria:

* 1.Signed informed consent from legal guardian of the subjects;
* Subjects are willing and able to cooperate to complete scheduled visits, treatment plans and laboratory tests and other procedures;
* Diagnosed as PWS by gene test;
* Age: 1 month (30 days after birth) - 5 years of age;
* Male or female;
* Calculated by Peabody Developmental Motor Scale, total motor quotient, gross motor quotient or fine motor quotient is less than 90 points;
* Thyroid function is within the normal reference range or remained within the normal reference range by substitution therapy;
* No history of rhGH therapy before.

Exclusion Criteria:

* Subjects with abnormal liver or kidney function;
* Subjects with obvious central sleep apnea and/or moderate or severe obstructive sleep apnea, acute lung infection;
* Subjects with chronic diseases that have long-term effects on bone metabolism and body composition;
* Subjects with congenital skeletal dysplasia, or spine scoliosis with moderate and above degree requiring treatment or lameness;
* Subjects with history of congenital heart disease, or an echocardiogram showing that the structural abnormalities require surgery or interventional therapy or that the left ventricular ejection fraction is <40%, or the abnormal electrocardiogram requiring intervention;
* Subjects with history of convulsions or epilepsy;
* Subjects with other systemic chronic diseases;
* Subjects with diagnosed tumors;
* Subjects with family history of cancers, a previous history of cancer, or considered to be a high risk of cancer combinating other information;
* Subjects with mental disease;
* Subjects with diabetes, or abnormal fasting glucose and researchers believe that may affect the safety of the subject;
* Subjects with severe obesity;
* Subjects with highly allergic constitution or allergy to proteins or investigational product or its excipient;
* Subjects who took part in other clinical trials within 3 months ;
* Subjects who received drug treatment that may interfere with GH secretion or GH action within 3 months;
* Other conditions in which the investigator preclude enrollment into the study

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-04-14 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
The change of the total motor quotient calculated by Peabody Developmental Motor Scale before and after treatment | Baseline, 26 weeks, 52 weeks

SECONDARY OUTCOMES:
Gross motor quotient and fine motor quotient calculated by Peabody Developmental Motor Scale before and after treatment | Baseline, 26 weeks, 52 weeks
Change of height standard deviation score (SDS) by chronological age before and after treatment | Baseline, 4 weeks, 13 weeks, 26 weeks, 39 weeks, 52 weeks
Body weight change before and after treatment | Baseline, 4 weeks, 13 weeks, 26 weeks, 39 weeks, 52 weeks
Change of BMI (Body mass index) standard deviation score before and after treatment | Baseline, 4 weeks, 13 weeks, 26 weeks, 39 weeks, 52 weeks
Global quotient, locomotor quotient, personal-social development quotient, language quotient, eye and hand coordination quotient, performance quotient and practical reasoning change calculated by Griffiths Mental Development Scale | Baseline, 26 weeks, 52 weeks
Bone maturation ( bone age/ chronological age: BA/CA) | Baseline, 52 weeks
Change of IGF-1(Insulin-like growth factor 1) SDS | Baseline, 4 weeks, 13 weeks, 26 weeks, 39 weeks, 52 weeks
IGF-1/IGFBP-3 molar ratio | Baseline, 4 weeks, 13 weeks, 26 weeks, 39 weeks, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Feihong Luo, Doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (6):
- China (6):
  - Tongji medical college huazhong university of science & technology, Wuhan, Hubei
  - The Children's Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Peking union medical college hospital, Beijing
  - Peking university first hospital, Beijing
  - Children's Hospital of Fudan University, Shanghai